CLINICAL TRIAL: NCT03266237
Title: Multi-parameter Immune Profile Associated With the Humoral Response to Influenza Vaccine, Vaxigrip® in Healthy and Frail Elderly Subjects Aged 65-90 Years in Singapore
Brief Title: The Immune Response to Influenza Vaccinations in Elderly Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); Agency for Science, Technology and Research (Other); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012/01214
Record Dates: First submitted 2016-09-20; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza; Influenza Virus Vaccines; Vaxigrip; Respiratory Tract Infections; Orthomyxoviridae Infections; Frailty; Aging; Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections; Orthomyxoviridae Infections; Frailty | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy Adult (Experimental): Healthy adult participants aged 21-40 years will be vaccinated with Vaxigrip® influenza vaccine
  Interventions: Drug: Vaxigrip®
- Healthy Elderly (Experimental): Healthy Elderly participants aged 65-90 years will be vaccinated with Vaxigrip® influenza vaccine.
  Interventions: Drug: Vaxigrip®
- Healthy Elderly Pre-Frail (Experimental): Healthy Elderly participants aged 65-90 years will be vaccinated with Vaxigrip® influenza vaccine.
  Interventions: Drug: Vaxigrip®
- Healthy Elderly Frail (Experimental): Healthy Elderly participants aged 65-90 years will be vaccinated with Vaxigrip® influenza vaccine.
  Interventions: Drug: Vaxigrip®

INTERVENTIONS:
Drug: Vaxigrip® — To describe the humoral immune response to Vaxigrip (IM) vaccination at Day 0 (baseline) and Day 28 according to the age and frailty status at baseline (i.e. in each study group) for each Influenza strain.

SUMMARY:
The aim of this study is to characterize the immune profile of frail and healthy aged individuals and investigate their immune responsiveness including the response to influenza vaccine over an 18-month period. The project will include a longitudinal study to define immune signatures and multi-parameter profiles associated with frailty and may lead to the identification of predictive markers of evolution to frailty and Immunosenescence in the elderly.

DETAILED DESCRIPTION:
With better healthcare available and improved accessibility, people are living longer. However, a majority of older persons cannot be considered to be aging well. Approximately 70% of those aged 85 years or older require frequent long hospitalizations because of their increased susceptibility to infections, cancers, dementia, and other age-related health problems, along with overall loss of function and autonomy associated with old age. Previous studies have shown that vaccination against influenza, which significantly reduces all-cause mortality in the elderly (65 years and older), was less immunogenic and effective with age. Frailty, a geriatric syndrome associated with low functional activity, weight loss, exhaustion, disability, decreased resilience to stressors, has been shown to increase risk for adverse outcomes and death. Better understanding the relationship between aging and waning immune responsiveness will enable the development of strategies to improve response to vaccination in the elderly and reduce morbidity and eventually mortality associated with age related complications and outcomes such as infectious diseases or frailty. A comprehensive analysis of the immune phenotype and function after antigenic challenge in older individuals would be a unique approach to understand (i) the potential associations between aging, impaired immune function and transition to frailty, (ii) which components of the immune system are altered with aging (innate vs adaptive immunity) and (iii) if early and/or late immune responses are preferentially altered with aging and frailty.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 65 years and <90 years on the day of inclusion for the elderly group, and ≥ 21-<40 for the adult group.
2. Informed consent form has been signed and dated.
3. Able to attend all scheduled visits and to comply with all trial procedures.
4. Living at home.
5. Able to walk without personal assistance and no other physical limitations that can limit participation.
6. Recruited from the cohort in Singapore Longitudinal Ageing Study-II (SLAS-II), as well as from sites in West Jurong and from Outpatient clinics at National University Hospital (NUH).

Exclusion Criteria:

1. Participation at the time of study enrollment (or in the 4 weeks preceding trial vaccination) or planned participation during the present trial period in another clinical trial investigating vaccine, drug, medical device, or medical procedure.
2. Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following trial vaccination, including influenza vaccination. However, 23-valent pneumococcal vaccine and tetanus vaccine will be allowed during this time window.
3. Receipt of an influenza vaccine within the 6 months preceding the trial vaccination or planned influenza vaccination during the trial.
4. Known or suspected congenital or acquired immunodeficiency or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
5. Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components or a history of a life-threatening reaction to Vaxigrip® or to a vaccine containing any of the same substances.
6. Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
7. Current alcohol or drug addiction.
8. Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
9. Identified as an Investigator or employee of the Investigator or study centre with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse) of the Investigator or employee with direct involvement in the proposed study.
10. Severe audio-visual impairment.
11. Dementia, severe cognitive impairment (MMSE <18), major depression or other psychotic disorders.
12. Progressive, degenerative neurologic disease: e.g. Alzheimer's disease.
13. Rapidly progressive or terminal illness under palliative care with life expectancy less than 12 months.
14. Primary severely muscle/joint disorders resulting in physical disability interfering with the physical performance tests needed for the study.
15. Hospital admission in the past 6 weeks.
16. (Relevant for the healthy young adults subjects group). Subject is pregnant (or positive urine pregnancy test), or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination).
17. Self-reported thrombocytopenia, contraindicating intramuscular vaccination
18. Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding vaccination, contraindicating intramuscular vaccination upon investigator's judgement.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The Immune Responsiveness of Elderly Subjects when Administered Influenza Vaccination as Measured by HAI | 18-month period
  Hemagglutination Inhibition (HAI) titer

SECONDARY OUTCOMES:
Cellular Immune Response and Inflammatory Profile of elderly subjects when administered influenza vaccination - Flu-Specific T cells | 18 months
  % Flu-specific T cells out of total PBMCs
Flu-Specific B Cell Response | 18 months
  No. of flu-specific B cells quantified out of 1x105 PBMCs
Inflammatory Markers | 18 months
  Quantitative (pg/mL analyte, picogram of analyte per milliliter of plasma)

OTHER OUTCOMES:
Clinical Assessments of the elderly subjects - Weight | 18 months
  Quantitative Weight (kg, kilograms)
Clinical Assessments of the elderly subjects - Height | 18 months
  Quantitative Height (m, meters)
Clinical Assessments of the elderly subjects - BMI | 18 months
  Quantitative BMI (weight and height will be combined to report in kg/m2)
Clinical Assessments of the elderly subjects - DXA | 18 months
  Quantitative Dual-Energy X-Ray Absorptiometry (DXA) scan: Standardized Muscle Index (appendicular lean mass / height-squared); T-score based on Bone Mineral Density BMD (appendicular lean mass and height will be combined to report in g/cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Paul Anantharajah Tambyah, MD, Principal Investigator — National University of Singapore
Locations (9):
- Singapore (9):
  - Moral Neighbourhood Link @ Telok Blangah, Singapore
  - National University Hospital, Singapore
  - THK Seniors Activity Centre @ Henderson (Satellite 93), Singapore
  - Moral Neighbourhood Link (Bukit Merah View), Singapore
  - THK Seniors Activity Centre @ Beo Crescent, Singapore
  - SARAH Senior Activity Centre, Singapore
  - THK Seniors Service @ Taman Jurong, Singapore
  - TaRa @ Jurong Point, Jurong West Central 2, Singapore
  - Outpatient Clinic, St Luke's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Publication of the data in peer-reviewed journals
Supporting Information: Study Protocol
Time Frame: five years approx
Access Criteria: through a research agreement

REFERENCES:
- [Derived] Camous X, Visan L, Ying CTT, Abel B, Nyunt MSZ, Narang V, Poidinger M, Carre C, Sesay S, Bosco N, Burdin N, Tambyah PA, Pin NT, Larbi A. Healthy elderly Singaporeans show no age-related humoral hyporesponsiveness nor diminished plasmablast generation in response to influenza vaccine. Immun Ageing. 2018 Nov 12;15:28. doi: 10.1186/s12979-018-0137-4. eCollection 2018. PMID 30455722